CLINICAL TRIAL: NCT03131479
Title: An Open-label, Parallel-group Study to Assess the Effect of LIK066 on Urinary Glucose Excretion, Pharmacokinetics, Safety and Tolerability Following Multiple Dose Administration in Patients With Decreased Renal Function Compared to Subjects With Normal Renal Function
Brief Title: Study of PK/PD, Safety and Tolerability of LIK066 in Patients With Decreased Renal Function.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLIK066B2202; 2016-004770-18 (EudraCT Number)
Record Dates: First submitted 2017-04-17; First posted 2017-04-27 (Actual); Results first posted 2019-02-06 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-06

CONDITIONS: Renal Impairment
Keywords: renal function; sodium-glucose co-transporter; pharmacokinetics; decreased renal function; decreased kidney function; kidney disease; urinary glucose excretion; UGE
MeSH Terms: conditions — Renal Insufficiency; Kidney Diseases | interventions — licogliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Mild (Experimental): Patients with mild renal impairment (Group 1) received LIK066 50 mg qd before breakfast for 7 days.
  Interventions: Drug: LIK066
- Moderate A (Experimental): Patients with moderate renal impairment grade A (Group 2) received LIK066 50 mg qd before breakfast for 7 days.
  Interventions: Drug: LIK066
- Moderate B (Experimental): Patients with moderate renal impairment grade B (Group 3) received LIK066 50 mg qd before breakfast for 7 days.
  Interventions: Drug: LIK066
- Severe (Experimental): Patients with severe renal impairment (Group 4) received LIK066 50 mg qd before breakfast for 7 days.
  Interventions: Drug: LIK066
- Normal (Experimental): Patients with normal renal function (Group 5) received LIK066 50 mg qd before breakfast for 7 days.
  Interventions: Drug: LIK066

INTERVENTIONS:
Drug: LIK066 — LIK066 50 mg tablets taken orally once daily before breakfast for 7 days.

SUMMARY:
The purpose of this trial was to evaluate whether the study drug, LIK066, causes glucose excretion in urine in patients with varying degrees of decreased kidney function and in subjects with normal kidney function. Blood samples were collected to measure the concentrations of LIK066 and to study the pharmacokinetics of LIK066. Pharmacokinetics is meant to study how LIK066 is absorbed, distributed and eliminated, in other words what the body does to the drug. The results of this study may be used to help determine whether LIK066 can be used to treat people with reduced kidney function and the proper dosing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.
* Male and female subjects age 18-78 years, inclusive, with controlled health condition as determined by past medical history, physical examination, electrocardiogram and laboratory test at screening.
* patients with Type 2 diabetes, HbA1c <10% at screening.
* Body mass index (BMI) ≤ 50 kg/m^2 at screening.

Exclusion Criteria:

* Patients with Type 1 diabetes
* Evidence of clinically significant liver function test: ALT, AST, gamma-GT, alkaline phosphatase >3 X ULN; serum bilirubin > 1.5 X ULN.
* Patients undergoing any method of dialysis
* clinically significant GI disorder related to malabsorption or that may affect drug or glucose absorption.
* subjects who experienced ketoacidosis, lactic acidosis or hyperosmolar coma within 6 months of screening visit.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=371

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 1 centers in the United States.
Period: Overall Study
Arm/Group | Mild | Moderate A | Moderate B | Severe | Normal
Started | 10 | 10 | 11 | 12 | 10
Safety Analysis Set (SS) (All subjects that received study drug) | 10 | 10 | 11 | 12 | 10
Pharmacokinetic Analysis Set (PAS) (At least one dose of study drug and had at least 1 valid PK concentration measurement) | 10 | 10 | 11 | 12 | 10
Pharcodynamic Analysis Set (PD) (At least one dose of study drug and had at least 1 valid post baseline PD) | 10 | 10 | 11 | 12 | 10
Completed | 10 | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 1 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0
Not completed — Subject/Guardian Decision | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mild | Moderate A | Moderate B | Severe | Normal | Total
Number analyzed (Participants) | 10 | 10 | 11 | 12 | 10 | 53
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.4 (9.03) | 66.3 (8.10) | 65.8 (9.10) | 63.3 (12.66) | 59.3 (8.17) | 64.0 (9.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 8 | 3 | 6 | 28
  Male | 4 | 5 | 3 | 9 | 4 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 3 | 1 | 3 | 3 | 4 | 14
  White | 7 | 9 | 8 | 9 | 5 | 38
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
24-hour Urinary glucose excretion (UGE) [Mean (Standard Deviation); unit: gram (g)] | 4.7 (9.96) | 2.9 (6.27) | 0.1 (0.12) | 0.3 (0.77) | 0.1 (0.07) | 1.5 (5.25)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 24-hour Urinary Glucose Excretion (UGE) on Day 7
Description: Urine was collected over 24 h to measure Urinary Glucose Excretion (UGE) at baseline (Day -1), following a single dose (Day 1) and at the end of the 7-day treatment (Day 7) to assess the effect of a 7 day treatment with LIK066 in subjects with decreased renal function compared to those with normal renal function.
Time Frame: Baseline , Day 7
Population: Pharmacodynamic Analysis Set (PD), which consisted of all participants with an observed PD value, was considered. Only patients with evaluable data at each time point were analyzed for that time point.
Measure: Mean (Standard Deviation); unit: gram (g)
Arm/Group | Normal | Mild | Moderate A | Moderate B | Severe
Number analyzed (Participants) | 10 | 10 | 10 | 11 | 12
gram (g) | 40.45 (21.93) | 31.87 (13.79) | 36.27 (19.51) | 19.88 (18.66) | 5.50 (3.75)
Statistical Analysis 1: Comparison: Normal vs Mild; Test type: Equivalence — Change from baseline was analyzed using a repeated measures model which included diabetic status, renal function, day and renal function*day and diabetic status*day as fixed factors and age, baseline body weight and baseline fasting plasma glucose as covariates; p = 0.154, Regression, Logistic; An unstructured variance-covariance structure was used. Baseline is defined to be the measurement collected on Day -1; adjusted arithmetic mean difference = -9.21, 90% CI 2-sided [-19.88 to 1.45]
Statistical Analysis 2: Comparison: Normal vs Moderate A; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.343, Regression, Logistic; adjusted arithmetic mean difference = -6.05, 90% CI 2-sided [-16.65 to 4.55]
Statistical Analysis 3: Comparison: Normal vs Moderate B; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.001, Regression, Logistic; adjusted arithmetic mean difference = -21.5, 90% CI 2-sided [-31.79 to 4.55]
Statistical Analysis 4: Comparison: Normal vs Severe; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.000, Regression, Logistic; adjusted arithmetic mean difference = -35.6, 90% CI 2-sided [-46.00 to -25.11]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for LIK066
Description: Plasma PK samples were collected at Day 1 and Day 7 and assayed for LIK066 concentrations using validated liquid chromatography-tandem mass spectrometry assays (LC MS/MS). The method will have an LLOQ of at least 5 ng/mL for LIK066. Concentrations were expressed in mass per volume units and refered to LIK066 plasma concentrations.
  Cmax was determined using the actual recorded sampling times and non-compartmental method(s) to assess the effect of a 7 day treatment with LIK066 in subjects with decreased renal function compared to those with normal renal function. Only descriptive analysis done.
Time Frame: Day 1 and Day 7 (0 hour predose and 0.5, 1.0, 2.0, 3.0, 4.0, 6.0, 8.0 and 12.0 hours post-dose)
Population: Pharmacokinetic Analysis Set (PAS), which consisted of all participants with at least 1 valid PK concentration measurement, was considered. Only patients with evaluable data at each time point were analyzed for that time point. Only descriptive analysis done.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Normal | Mild | Moderate A | Moderate B | Severe
Number analyzed (Participants) | 10 | 10 | 10 | 11 | 12
nanogram per milliliter (ng/mL)
  Day 1 | 565 (176) | 590 (176) | 492 (142) | 569 (147) | 650 (199)
  Day 7: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
  Day 7 | 650 (250) | 678 (219) | 686 (243) | 743 (301) | 800 (268)

3. Primary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) for LIK066
Description: Plasma PK samples were collected at Day 1 and Day 7 and assayed for LIK066 concentrations using validated liquid chromatography-tandem mass spectrometry assays (LC MS/MS). The method will have an LLOQ of at least 5 ng/mL for LIK066. Concentrations were expressed in mass per volume units and refered to LIK066 plasma concentrations.
  Tmax was determined using the actual recorded sampling times and non-compartmental method(s) to assess the effect of a 7 day treatment with LIK066 in subjects with decreased renal function compared to those with normal renal function. Only descriptive analysis done.
Time Frame: Day 1 and Day 7 (0 hour predose and 0.5, 1.0, 2.0, 3.0, 4.0, 6.0, 8.0 and 12.0 hours post-dose)
Population: as for outcome 2
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | Normal | Mild | Moderate A | Moderate B | Severe
Number analyzed (Participants) | 10 | 10 | 10 | 11 | 12
hour (hr)
  Day 1 | 1.00 [0.500 to 4.03] | 1.00 [0.500 to 4.00] | 1.00 [1.00 to 8.00] | 1.00 [0.500 to 3.00] | 1.00 [0.500 to 4.00]
  Day 7: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
  Day 7 | 1.00 [0.500 to 3.00] | 1.03 [0.500 to 4.00] | 1.00 [0.500 to 6.00] | 1.00 [0.500 to 2.00] | 1.00 [0.500 to 2.00]

4. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the End of the Dosing Interval Tau (AUCtau) for LIK066
Description: Plasma PK samples were collected at Day 1 and Day 7 and assayed for LIK066 concentrations using validated liquid chromatography-tandem mass spectrometry assays (LC MS/MS). The method will have an LLOQ of at least 5 ng/mL for LIK066. Concentrations were expressed in mass per volume units and refered to LIK066 plasma concentrations.
  AUCtau was determined using the actual recorded sampling times and non-compartmental method(s) to assess the effect of a 7 day treatment with LIK066 in subjects with decreased renal function compared to those with normal renal function. Only descriptive analysis done.
Time Frame: Day 1 and Day 7 (0 hour predose and 0.5, 1.0, 2.0, 3.0, 4.0, 6.0, 8.0 and 12.0 hours post-dose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (hr*ng/mL)
Arm/Group | Normal | Mild | Moderate A | Moderate B | Severe
Number analyzed (Participants) | 10 | 10 | 10 | 11 | 12
hour*nanogram per milliliter (hr*ng/mL)
  Day 1: number analyzed (Participants) | 10 | 10 | 9 | 11 | 12
  Day 1 | 2830 (650) | 3330 (563) | 3120 (567) | 3360 (886) | 4150 (1040)
  Day 7: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
  Day 7 | 3440 (790) | 4170 (981) | 4080 (1040) | 4510 (1240) | 6290 (2280)

5. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) for LIK066 on Day 7
Description: Plasma PK samples were collected at Day 1 and Day 7 and assayed for LIK066 concentrations using validated liquid chromatography-tandem mass spectrometry assays (LC MS/MS). The method will have an LLOQ of at least 5 ng/mL for LIK066. Concentrations were expressed in mass per volume units and refered to LIK066 plasma concentrations.
  AUClast was determined using the actual recorded sampling times and non-compartmental method(s) to assess the effect of a 7 day treatment with LIK066 in subjects with decreased renal function compared to those with normal renal function. AUClast is similar to AUCtau on Day 1 since the Tlast for Day 1 = 24hrs (tau = 24hrs); therefore AUClast is not reported for Day1, it is however reported for Day 7 since the Tlast is different from 24 hours. Only descriptive analysis done.
Time Frame: Day 7 (0 hour predose and 0.5, 1.0, 2.0, 3.0, 4.0, 6.0, 8.0 and 12.0 hours post-dose)
Population: Pharmacokinetic Analysis Set (PAS), which consisted of all participants with at least 1 valid PK concentration measurement, was considered. Only descriptive analysis done.
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (hr*ng/mL)
Arm/Group | Normal | Mild | Moderate A | Moderate B | Severe
Number analyzed (Participants) | 10 | 10 | 10 | 11 | 12
hour*nanogram per milliliter (hr*ng/mL) | 4190 (1090) | 5280 (1540) | 5440 (1740) | 6410 (2160) | 9620 (3910)

6. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUCinf) for LIK066 on Day 1
Description: Plasma PK samples were collected at Day 1 and Day 7 and assayed for LIK066 concentrations using validated liquid chromatography-tandem mass spectrometry assays (LC MS/MS). The method will have an LLOQ of at least 5 ng/mL for LIK066. Concentrations were expressed in mass per volume units and refered to LIK066 plasma concentrations.
  AUCinf was determined using the actual recorded sampling times and non-compartmental method(s) to assess the effect of a 7 day treatment with LIK066 in subjects with decreased renal function compared to those with normal renal function. AUCinf is a single dose parameter and therefore is presented on Day 1 only, after the first dose of LIK066. Only descriptive analysis done.
Time Frame: Day 1 (0 hour predose and 0.5, 1.0, 2.0, 3.0, 4.0, 6.0, 8.0 and 12.0 hours post-dose)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (hr*ng/mL)
Arm/Group | Normal | Mild | Moderate A | Moderate B | Severe
Number analyzed (Participants) | 10 | 10 | 10 | 11 | 12
hour*nanogram per milliliter (hr*ng/mL) | 310 (688) | 3610 (649) | 3440 (551) | 3520 (1000) | 4450 (1480)

7. Primary Outcome: Terminal Elimination Half-life (T1/2) for LIK066 on Day 7
Description: Plasma PK samples were collected at Day 1 and Day 7 and assayed for LIK066 concentrations using validated liquid chromatography-tandem mass spectrometry assays (LC MS/MS). The method will have an LLOQ of at least 5 ng/mL for LIK066. Concentrations were expressed in mass per volume units and refered to LIK066 plasma concentrations.
  T1/2 was determined using the actual recorded sampling times and non-compartmental method(s) to assess the effect of a 7 day treatment with LIK066 in subjects with decreased renal function compared to those with normal renal function. T1/2 is only reported at Day 7 only, since there was sampling out to ~5 half-lives after the Day 7 dose of LIK066. Only descriptive analysis done.
Time Frame: Day 7 (0 hour predose and 0.5, 1.0, 2.0, 3.0, 4.0, 6.0, 8.0 and 12.0 hours post-dose)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hour (hr)
Arm/Group | Normal | Mild | Moderate A | Moderate B | Severe
Number analyzed (Participants) | 10 | 10 | 10 | 11 | 12
hour (hr) | 22.9 (20.3) | 21.8 (10.8) | 21.1 (9.25) | 20.9 (8.91) | 22.8 (9.52)

8. Primary Outcome: Apparent Systemic (or Total Body) Clearance From Plasma Following Extravascular Administration (CL/F) for LIK066 on Day 1
Description: Plasma PK samples were collected at Day 1 and Day 7 and assayed for LIK066 concentrations using validated liquid chromatography-tandem mass spectrometry assays (LC MS/MS). The method will have an LLOQ of at least 5 ng/mL for LIK066. Concentrations were expressed in mass per volume units and refered to LIK066 plasma concentrations.
  CL/F was determined using the actual recorded sampling times and non-compartmental method(s) to assess the effect of a 7 day treatment with LIK066 in subjects with decreased renal function compared to those with normal renal function. Since Day 7 represented steady state of LIK066 in the study, the appropriately calculated steady-state clearance parameter computed was CLss/F and was presented. Only descriptive analysis done.
Time Frame: Day 1 (0 hour predose and 0.5, 1.0, 2.0, 3.0, 4.0, 6.0, 8.0 and 12.0 hours post-dose)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Liter per hour (L/h)
Arm/Group | Normal | Mild | Moderate A | Moderate B | Severe
Number analyzed (Participants) | 10 | 10 | 10 | 11 | 12
Liter per hour (L/h) | 17.4 (4.20) | 14.3 (2.59) | 14.9 (2.55) | 15.4 (4.87) | 12.4 (4.53)

9. Primary Outcome: Apparent Volume of Distribution During the Terminal Elimination Phase Following Extravascular Administration (Vz/F) for LIK066 on Day 1
Description: Plasma PK samples were collected at Day 1 and Day 7 and assayed for LIK066 concentrations using validated liquid chromatography-tandem mass spectrometry assays (LC MS/MS). The method will have an LLOQ of at least 5 ng/mL for LIK066. Concentrations were expressed in mass per volume units and refered to LIK066 plasma concentrations.
  Vz/F was determined using the actual recorded sampling times and non-compartmental method(s) to assess the effect of a 7 day treatment with LIK066 in subjects with decreased renal function compared to those with normal renal function. Only descriptive analysis done.
Time Frame: Day 1 (0 hour predose and 0.5, 1.0, 2.0, 3.0, 4.0, 6.0, 8.0 and 12.0 hours post-dose)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Liter (L)
Arm/Group | Normal | Mild | Moderate A | Moderate B | Severe
Number analyzed (Participants) | 10 | 10 | 10 | 11 | 12
Liter (L) | 160 (59.4) | 140 (28.6) | 164 (79.9) | 176 (67.8) | 134 (50.5)

10. Primary Outcome: Renal Clearance From Plasma (CLr) for LIK066
Description: Urine PK samples were collected at Day 1 and Day 7 and assayed for LIK066 concentrations using validated liquid chromatography-tandem mass spectrometry assays (LC MS/MS). The method will have an LLOQ of at least 5 ng/mL for LIK066. Concentrations were expressed in mass per volume units and refered to LIK066 plasma concentrations.
  CLr was determined using the actual recorded sampling times and non-compartmental method(s) to assess the effect of a 7 day treatment with LIK066 in subjects with decreased renal function compared to those with normal renal function. Only descriptive analysis done.
Time Frame: Day 1 and Day 7 (0 hour predose and 0.5, 1.0, 2.0, 3.0, 4.0, 6.0, 8.0 and 12.0 hours post-dose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liter per hour (L/hr)
Arm/Group | Normal | Mild | Moderate A | Moderate B | Severe
Number analyzed (Participants) | 10 | 10 | 10 | 11 | 12
Liter per hour (L/hr)
  Day 1: number analyzed (Participants) | 10 | 10 | 9 | 11 | 12
  Day 1 | 0.389 (0.179) | 0.348 (0.141) | 0.259 (0.114) | 0.173 (0.0919) | 0.0522 (0.0237)
  Day 7: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
  Day 7 | 0.474 (0.275) | 0.367 (0.0815) | 0.294 (0.119) | 0.174 (0.0636) | 0.0694 (0.0461)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 7 months
Arm/Group | Normal | Mild | Moderate A | Moderate B | Severe
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 1/11 | 1/12
Other Adverse Events (participants affected / at risk) | 9/10 | 10/10 | 10/10 | 11/11 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normal (N=10) | Mild (N=10) | Moderate A (N=10) | Moderate B (N=11) | Severe (N=12)
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Normal (N=10) | Mild (N=10) | Moderate A (N=10) | Moderate B (N=11) | Severe (N=12)
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 1 | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 9 | 10 | 10 | 10 | 11
Flatulence (Gastrointestinal disorders) | 7 | 7 | 6 | 9 | 7
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-01-11): https://cdn.clinicaltrials.gov/large-docs/79/NCT03131479/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/79/NCT03131479/SAP_001.pdf